CLINICAL TRIAL: NCT07234019
Title: A Randomized, Open-label Study To Compare The Efficacy And Safety Of Rituximab Combining Anti-CD38 Monoclonal Antibody Versus Rituximab in ITP Patients Who Failed or Relapsed After Glucocorticoid Therapy
Brief Title: Rituximab Combining Anti-CD38 Monoclonal Antibody Versus Rituximab in the Management of Primary Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023053
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rituximab combined with Daratumumab（anti-CD38 monoclonal antibody） (Experimental): Rituximab (375mg/m2) was given once (day1) and a Daratumumab (16mg/kg) was given four times (day8,15,22,29).
  Interventions: Drug: Daratumumab（Anti-CD38 Monoclonal Antibody）; Drug: Rituximab
- rituximab (Active Comparator): Rituximab (375mg/m2) was given once.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Daratumumab（Anti-CD38 Monoclonal Antibody） — All subjects were randomly assigned to group A (active comparator) and group B (experimental). For subjects in group B (experimental), rituximab (375mg/m2) was given once (day1) and Daratumumab (16mg/kg) was given four times (day8,15,22,29).
  Arms: rituximab combined with Daratumumab（anti-CD38 monoclonal antibody）
Drug: Rituximab — All subjects were randomly assigned to group A (active comparator) and group B (experimental). For subjects in group A (active comparator) , rituximab (375mg/m2) was given once. For subjects in group B (experimental), rituximab (375mg/m2) was given once (day1) and anti-CD38 monoclonal antibody (16mg/kg) was given four times (day8,15,22,29).

SUMMARY:
This randomized, open-label study aim to compare the efficacy and safety of rituximab combining anti-CD38 monoclonal antibody with rituximab in ITP patients.This study will be conducted in ITP patients who had not responded to or had relapsed after previous glucocorticoid treatment.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for recurrent and refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.

The main pathogenesis of ITP is the loss of platelet autoantigen immune tolerance, which leads to abnormal activation of humoral and cellular immunity. It is characterized by antibody mediated platelet destruction and insufficient platelet production by megakaryocytes. The residual long-term autoreactive plasma cells may be a source of therapeutic resistance to autoimmune cytopenia. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. Therefore, the strategy of simply eliminating B cells may not work, because LLPC will continue to produce pathogenic antibodies. In view of this, the investigators expected that the combination of rituximab and anti-CD38 monoclonal antibody could simultaneously eliminate CD20 positive B cells and LLPC, thereby profoundly reducing the production of pathogenic antibodies and increasing the efficacy of ITP treatment. Some patients have been treated with this regimen in the past, with good efficacy and safety. Therefore, the investigators planned to conduct a clinical study to evaluate the safety and efficacy of rituximab combined with Daratumumab（anti-CD38 monoclonal antibody）versus rituximab in relapsed adult patients with primary immune thrombocytopenia, in order to provide more treatment options for patients with ITP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female.
* Before enrollment, the subjects have been clinically diagnosed with primary immune thrombocytopenia for no less than three months according to the American Society of Hematology guidelines 2011 Evidence-Based Practice Guideline (Neunert et al. 2011) or the International Consensus Report for the Investigation and Management of Primary Immune Thrombocytopenia (Provan et al. 2010), as applicable locally.
* Subjects with a platelet count of <30×10^9/L within the 48 hours prior to the first dose of the study drug;The platelet count of at least two separate assessments (at least 1 week apart) <30×10^9/L during the screening visit.
* Patients have failed glucocorticoid therapy (either due to inefficacy, efficacy could not be maintained, or relapse).
* Previous emergency treatment for ITP (e.g., methylprednisolone, platelet, gamma globulin infusion) must have been completed at least 2 weeks before the first dose.
* Hepatic and renal function (e.g., alanine aminotransferase, aspartate aminotransferase, total bilirubin, serum creatinine) <1.5 times the upper limit of normal (ULN).
* ECOG performance status score of ≤2.
* Cardiac function: New York Heart Association (NYHA) class ≤2.
* Enrollment of subjects receiving maintenance therapy is permitted, including glucocorticoids (≤0.5 mg/kg of prednisone or equivalent) or TPO receptor agonists, but the concomitant medication must have been stable for a minimum of 4 weeks prior to the initial infusion of the study drug; Azathioprine, danazol, cyclosporine A, tacrolimus, sirolimus, etc. must be stopped at least 4 weeks before the first dose; CD20 monoclonal antibody such as rituximab must have been stopped for more than 6 months; the interval between splenectomy and first administration need to be more than 6 months.
* For fertile female patients, a negative pregnancy test result is required. Fertile female and male patients must use effective contraception separately during the study and for 90 days after the cessation of study drug treatment.
* Subjects comprehensively understand and can adhere to the study protocol requirements and willingly signed the informed consent form.

Exclusion Criteria:

* Uncontrollable primary diseases of important organs, such as malignant tumors, liver failure, heart failure, renal failure and other diseases.
* HIV positive.
* Accompanied by uncontrollable active infection, including hepatitis B, hepatitis C, cytomegalovirus, EB virus and syphilis positive.
* Accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage, etc..
* At present, there are heart diseases, arrhythmias that need treatment or hypertension that researchers judge is poorly controlled.
* Patients with thrombotic diseases such as pulmonary embolism, thrombosis and atherosclerosis.
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past.
* atients with mental disorders who cannot normally obtain informed consent and conduct trials and follow-up.
* Patients whose toxic symptoms caused by pre-trial treatment have not disappeared.
* Other serious diseases that may limit the subject's participation in this test (such as diabetes; Severe cardiac insufficiency; Myocardial obstruction or unstable arrhythmia or unstable angina pectoris in recent 6 months; Gastric ulcer, etc.).
* Patients with septicemia or other irregular severe bleeding.
* Patients taking antiplatelet drugs at the same time.
* Pregnant women, suspected pregnancies (positive pregnancy test for human chorionic gonadotropin in urine at screening) and lactating patients.
* Subjects with a known allergy to medications were used in the trial or excipients.
* Any other conditions unsuitable for participation in this study, as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate at week 12 | 12 weeks
  Overall response rate was defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding and subjects with a platelet count ≥ 100 × 10^9/L without bleeding at week 12 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.

SECONDARY OUTCOMES:
Complete remission rate at week 12 | 12 weeks
  Complete remission rate was defined as proportion of subjects with a platelet count ≥ 100 × 10^9/L without bleeding at week 12 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.
Partial remission rate at week 12 | 12 weeks
  Partial remission rate was defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding at week 12 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.
Overall response rate at month 6 | 6 months
  Overall response rate was defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding and subjects with a platelet count ≥ 100 × 10^9/L without bleeding at month 6 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.
Overall response rate at month 12 | 12 months
  Overall response rate was defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding and subjects with a platelet count ≥ 100 × 10^9/L without bleeding at month 12 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.
Sustained response rate at month 6 | 6 months
  Proportion of subjects who keep a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding and subjects who keep a platelet count ≥ 100 × 10^9/L without bleeding at month 6 after initial administration.
Sustained response rate at month 12 | 12 months
  Proportion of subjects who keep a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding and subjects who keep a platelet count ≥ 100 × 10^9/L without bleeding at month 12 after initial administration.
Time to response (TTR) | 12 months
  Time needed from treatment initiation to platelet count ≥30×10^9/L and at least twice the baseline platelet count.
Maintenance time | 12 months
  Time from response to relapse.
Rescue treatment | 12 weeks
  Percentage of patients who need rescue treatment within 12 weeks during the study period.
Concomitant maintenance drug | 12 weeks
  Changes in concomitant maintenance therapy at week12 compared with that before the study.
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale | 12 weeks
  Changes of the subjects' numbers in WHO bleeding score after treatment according to the reported World Health Organization's Bleeding Scale at week 12. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Adverse events assessment | 12 months
  Incidence, severity, and relationship of treatment emergent adverse events during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI